CLINICAL TRIAL: NCT06417697
Title: A Phase 1b, Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Effects of XEN-101 on Safety, Tolerability, and Pharmacodynamics in Subjects with Obesity
Brief Title: A Phase 1b Study to Evaluate the Safety of XEN-101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study not stopped for safety reasons. Data were reviewed after the first 23 patients had completed scheduled dosing and there was no signal of efficacy for change in body weight. This clinical trial has been determined to be futile.
Sponsor: Xeno Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XB-101-102
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XEN-101 (Experimental)
  Interventions: Drug: XEN-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN-101 — capsule formulation
  Arms: XEN-101
Drug: Placebo — capsule formulation
  Arms: Placebo

SUMMARY:
This Phase 1b study will evaluate the effects of XEN-101 in subjects with obesity

DETAILED DESCRIPTION:
This study will assess the safety, tolerability and weight loss associated with XEN-101 in obese men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 60 years, inclusive, at Screening
2. Body mass index of 30 to 45 kg/m2
3. Stable body weight for at least 3 months (i.e., fluctuation of ≤5%)
4. If a female of childbearing potential, must agree to use double barrier contraception (e.g., condom and 1 additional form of adequate contraception) from the date of signing of the ICF, throughout the study, and for 4 weeks after the final dose of study drug. In addition, she must be advised not to donate ova during this period. If a non-sterilized male is sexually active with a female partner of childbearing potential, he must use double barrier contraception from the date of signing of the ICF, throughout the study, and for 8 weeks after the final dose of study drug. In addition, he must be advised not to donate sperm during this period
5. If a female of childbearing potential, must have a negative pregnancy test at Screening and on Day 1 (baseline)
6. Able to provide informed consent
7. Willing and able to comply with this protocol and procedures, including feces collection, and be available for the entire duration of the study

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug study, or less than 30 days or 5 times the half-life of the drug candidate (whichever is longer) has passed between Screening for this study and the end of the Treatment Period of the previous investigational device or drug study
2. Diagnosed with type 1 diabetes or type 2 diabetes (T2D) (resolution of T2D >3 years before Screening is allowed)
3. Laboratory evidence during Screening of T2D, including glycated hemoglobin (HbA1c) ≥6.5% or fasting glucose ≥126 mg/dL (≥7.0 mmol/L)
4. Evidence of clinically significant cardiac, neurologic, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, or gastrointestinal disease that, in the Investigator's opinion, would compromise the safety of the subject, interfere with the interpretation of the study results, or otherwise preclude subject participation
5. Female who is pregnant, nursing, or intends to become pregnant during the study.
6. Positive result for hepatitis B virus surface antigen, hepatitis C virus ribonucleic acid, and human immunodeficiency virus (HIV) antibody at Screening
7. Use of anti-obesity medications (e.g., glucagon-like peptide-1 analogues, stimulants, bupropion/naltrexone) within 6 months before Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) | Day 1 through Day 43
  Assessing the type and frequency of adverse events
Effect on body weight | Day 1 through Day 43
  change and percent change from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No